CLINICAL TRIAL: NCT00412139
Title: A Correlation Between Histological Findings of the Blood Vessels in Patients With Chronic Renal Failure and Serum Uremic Toxins and Its Diagnostic Performance in the Assessment of the Cardiovascular Morbidity and Mortality
Brief Title: Serum Uremic Toxins and Histological Findings of the Blood Vessels in Dialysis Patients
Status: Completed | Type: Observational
Sponsor: University of Skopje (Other)
Collaborators: Ministry of Science and Education, R. Macedonia (Unknown)
Responsible Party: Goce Spasovski, PI, Department of Nephrology, University Clinical Center
Other Study IDs: 13-1001/2-05
Record Dates: First submitted 2006-12-12; First posted 2006-12-15 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2008-12

CONDITIONS: Chronic Renal Failure
Keywords: vascular calcifications; uremic toxins; renal osteodystrophy; Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Vascular Calcification; Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: None Retained — 3 aliquots of 2-3 ml sera are retained for various uremic markers determination
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients treated by chronic renal replacement therapy are exposed to cardiovascular problems and suffer from an accelerated and sever atherosclerosis. Classical risk factors for atherosclerosis and cardiovascular diseases (CVD) do not explain the full risk of CVD in the dialysis patients. Additional risk factors are therefore likely to exist. The uremic syndrome is attributed to the progressive retention of a large number of compounds, which under normal conditions are excreted by the healthy kidneys. Uremic toxins such are parathormone (PTH), vitamin D and phosphates, cause development of renal osteodystrophy (ROD), i.e. disordered calcium and phosphate metabolism. Both conditions of hyperparathyroid and adynamic bone disease (ABD) lead to an elevated calcium x phosphate product and increased vascular calcification, which might occur in intimal and medial layer of the vessel wall. It is important to consider these processes separately, as the vascular consequences (occlusion with atheromatosis and vascular stiffening through medial calcification) are different. Moreover, the difference between uremic and non-uremic intimal plaque is not the size but its composition, with markedly increased calcium content. Hence, these observations have an important socio-economic impact because of the increased cardiovascular morbidity and mortality.

The investigators hypothesized that uremic toxins in dialysis patients influence directly and/or indirectly the development of atherosclerosis, vascular calcifications and CVD.

DETAILED DESCRIPTION:
Rationale: Patients treated by chronic renal replacement therapy are exposed to cardiovascular problems and suffer from an accelerated and sever atherosclerosis. Classical risk factors for atherosclerosis and cardiovascular diseases (CVD) do not explain the full risk of CVD in the dialysis patients. Additional risk factors are therefore likely to exist. The uremic syndrome is attributed to the progressive retention of a large number of compounds, which under normal conditions are excreted by the healthy kidneys. Uremic toxins such are parathormone (PTH), vitamin D and phosphates, cause development of renal osteodystrophy (ROD), i.e. disordered calcium and phosphate metabolism. Both conditions of hyperparathyroid and adynamic bone disease (ABD) lead to an elevated calcium x phosphate product and increased vascular calcification, which might occur in intimal and medial layer of the vessel wall. It is important to consider these processes separately, as the vascular consequences (occlusion with atheromatosis and vascular stiffening through medial calcification) are different. Moreover, the difference between uremic and non-uremic intimal plaque is not the size but its composition, with markedly increased calcium content. Hence, these observations have an important socio-economic impact because of the increased cardiovascular morbidity and mortality.

Hypothesis: We hypothesized that uremic toxins in dialysis patients influence directly and/or indirectly the development of atherosclerosis, vascular calcifications and CVD.

Objectives:

To asses the histology of arterial vessels in patients with end-stage renal failure and to evaluate its relationship with serum uremic toxins.

To determine the biochemical and clinical risk factors that might influence the development of vascular calcifications and their diagnostic performance in the assessment of CVD morbidity and mortality.

Methods: A cross-sectional study will be conducted at the Department of Nephrology Skopje. After the initial assessment patients will be followed for 2 years as the prospective part of the study.

Seventy-five to ninety patients will be included, during one-year period or until proposed number of patients is recruited. The study cohort will be divided to 3 subgroups: 1) patients at the initiation of dialysis therapy, 2) patients on regular dialysis treatment for a few years and 3) patients undergoing renal transplantation. During the follow-up period cardiovascular and cerebrovascular events and the moment of their occurrence will be recorded, as well as the peripheral vascular diseases. Moreover, clinical, laboratory data and arterial vessel samples for histology will be collected at the moment of inclusion.

Expected outcomes: We expect the determination of high correlation coefficient between histological parameters and various uremic toxins, which are responsible for development atherosclerosis and vascular calcifications, leading to an accelerated progression of CVD in dialysis patients. This determination could help to design new preventive therapeutic tools in these patients. The result of this work will impose a positive impact on quality of life and therapeutic costs related to atherosclerosis not only in the dialysis populations but also in the pre-dialysis chronic renal failure populations and kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal failure patients with a need for creation of AV fistula
* Dialysis patients with a need of reanastomosing of the AV fistula (thrombosis or insufficient blood flow)

Exclusion Criteria:

* Diabetes
* Malignant disease
* Prior treatment with corticosteroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CKD patients with a need for dialysis within a few months CKD patients on dialysis with thormbosis of AV fistula CKD patients on dialysis scheduled for kidney transplantation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-12; Primary Completion 2008-11 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Goce Spasovski, MD, PhD, Principal Investigator — Department of Nephrology, University Clinical Center, Vodnjanska 17, 1000 Skopje, R. Macedonia; Momir Polenakovic, MD, PhD, Study Chair — Macedonian Academy of Science and Arts
Locations (1):
- Department of Nephrology, University Clinical Center, Skopje, North Macedonia